CLINICAL TRIAL: NCT03884751
Title: A Phase I Clinical Study of Chimeric Antigen Receptor T Cells Targeting Glypican-3 (CAR-GPC3 T Cells) in Patients With Advanced Hepatocellular Carcinoma
Brief Title: Chimeric Antigen Receptor T Cells Targeting Glypican-3
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CARsgen Therapeutics Co., Ltd. (Industry)
Collaborators: NanJing PLA 81 Hospital (Other); First Affiliated Hospital of Zhejiang University (Other); RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT011-HCC-01
Record Dates: First submitted 2019-02-25; First posted 2019-03-21 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; CAR-T
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-GPC3 T Cells (Experimental): The subjects are enrolled into 2 dose levels cohorts in sequence
  Interventions: Biological: CAR-GPC3 T Cells

INTERVENTIONS:
Biological: CAR-GPC3 T Cells — CAR-GPC3 T Cells injection
  Other Names: Chimeric Antigen Receptor T Cells Targeting Glypican-3

SUMMARY:
A Phase I Clinical Study of Chimeric Antigen Receptor T Cells Targeting Glypican-3 (CAR-GPC3 T Cells) in Patients with Advanced Hepatocellular Carcinoma

DETAILED DESCRIPTION:
This is a phase I open-label, single-arm, multicenter clinical trial designed to observe and evaluate the safety, cell metabolokinetics, and efficacy of CAR-GPC3 T cells infused intravenously at single escalating doses in patients with advanced hepatocellular carcinoma.

Primary objectives:

- To evaluate the safety and tolerability of CAR-GPC3 T cells infused intravenously at escalating doses in patients with advanced hepatocellular carcinoma.

Secondary objectives：

* To evaluate the metabolic kinetics of single infusion of CAR-GPC3 T cells
* To evaluate the overall safety and tolerability of infusion of CAR-GPC3 T cells
* To observe the efficacy of CAR-GPC3 T cells in the treatment of advanced hepatocellular carcinoma

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 70 years, male or female;
2. Patients with advanced hepatocellular carcinoma (HCC) diagnosed by histopathology or cytology who are not suitable for surgery or local treatment (including ablation, intervention, and radiotherapy), have developed progressive disease or intolerability after standard systemic therapies (including but not limited to systemic chemotherapy, molecular targeted therapy) and have no effective treatment at the time of enrollment;
3. According to RECIST 1.1, patients have at least one evaluable target lesion, defined as: the longest diameter of non-lymph node lesion ≥ 10 mm, or the shortest diameter of lymph node lesion ≥ 15 mm); hepatic lesions require arterial phase contrast enhancement;
4. In tumor tissue samples GPC3 is detected positive by immunohistochemistry (IHC);
5. According to Barcelona Clinic Liver Cancer staging(BCLC), the patients are classified into Grade C or Grade B unsuitable for local treatment/progressive disease after local treatment;
6. Expected survival is > 12 weeks;
7. Cirrhosis status Child-Pugh score: Grade A;
8. Eastern Cooperative Oncology Group(ECOG) Performance Status score: 0 to 1 point;
9. Without active hepatitis B and/or Hepatitis C;
10. Have venous accesses for pheresis;
11. Acceptable routine blood test showing no contraindication to the lymphodepletion pretreatment;
12. Adequate liver, renal, cardiovascular, respiratory function;
13. Subjects of childbearing age must undergo a serum pregnancy test within 14 days before the initiation of the study and the result must be negative. In addition, they should be willing to use a reliable method of contraception during the trial (within 24 months (M24) after cell infusion); male subjects whose spouses are women of childbearing age should undergo sterilization surgery or agree to use a reliable method of contraception during the trial;
14. Understand and sign informed consent.

Exclusion Criteria:

1. Pregnant or breast-feeding women;
2. HCV-RNA(Hepatitis C Virus RNA ), HIV antibodies or Syphilis Serological tests are positive;
3. HBV（Hepatitis B） and HCV(Hepatitis C virus ) infection exist simultaneously;
4. Any uncontrollable active infection
5. Patients who had received systemic steroids or other immunosuppressive agents
6. Previous or present hepatic encephalopathy;
7. Current clinically significant ascites;
8. ≥50% of the liver is replaced by tumor or portal vein main tumor thrombus, or tumor thrombus invasion of mesenteric vein / inferior vena cava;
9. Metastases to the central nervous system and clinically significant central nervous system diseases;
10. Patients with existing heart disease in need of treatment or hypertension that be poorly controlled
11. Patients with known active autoimmune diseases which require to be treated with immunosuppressive agents including biological agents;
12. Patients with a history of organ transplantation or waiting for organ transplantation (including liver transplantation);
13. Patients with local treatments such as surgical treatment, interventional therapy, radiotherapy, ablation or systemic chemotherapy were performed for the studied disease within 2 weeks prior to apheresis;Or received immunotherapy (PD-1/ PD-L1 monoclonal antibody, see Section 15) or any Chinese herbal or proprietary medicine for the control of liver cancer within 1 week prior to apheresis;Or received sorafenib, regofenib, ramvastinib and other tyrosine kinase inhibitor targeted drugs within 1 week prior to apheresis;Targeted therapy with anti-angiogenic monoclonal antibodies such as bevacizumab or its analogue 4 weeks prior to apheresis;
14. Patiens with previous treatment with targeted GPC3, TCR-T or CAR-T;
15. Patients who previously received anti-PD-1/ PD-L1 monoclonal antibody therapy within 4 weeks prior to apheresis;
16. Patients who had uncured malignant tumors in the past 5 years or at the same time, excluding in situ cervical cancer and skin basal cell carcinoma;
17. Other serious illnesses that may limit subjects to participate in the trial (such as poorly controlled diabetes mellitus, severe cardiac insufficiency , myocardial infarction or unstable arrhythmia or unstable angina pectoris within the last 6 months, lung embolism, chronic obstructive pulmonary diseases, interstitial pulmonary diseases,gastric ulcer, a history of gastrointestinal bleeding or a clear tendency to gastrointestinal bleeding;
18. According to the investigators' evaluation, patients are unable or unwilling to comply with the requirements of the study protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2021-12-03 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | After 28 days of single infusion
  Safety
Maximum tolerated dose (MTD) | After 28 days of single infusion
  tolerability

SECONDARY OUTCOMES:
Pharmacokinetics (the copies of cells in vivo) | Day0~Week 26
  Pharmacokinetics is the"Implantation endpoint" which is defined as the number of copies of CAR-GPC3 DNA in peripheral blood at each visit after infusion until any two consecutive test results are negative or below the detection limit. It aims to calculate the Peak Plasma Concentration (Cmax)
Pharmacokinetics ( the duration of survival of cells in vivo) | Day0~Week 26
  Duration of CAR-GPC3 T cell persistence is the period from the day of infusion to the first negative test result or result lower than the detection limit.It aims to calculate the area under the plasma concentration versus time curve (AUC)
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Month 24
  Adverse events up to 24 months of follow-up visit judged by the investigator to be associated with CAR-GPC3T cell infusion, such as abnormalities or changes in laboratory examinations, physical examinations, vital signs, etc.
Antitumor efficacy-Progression-free survival (PFS) | Month 24
  The period from the day when the subject receives the infusion of cells to the first recorded tumor progression (whether treated or not) or death of any cause, which occurs first.
Antitumor efficacy-Duration of response (DOR) | Month 24
  The period from the first evaluation of CR or PR to the first evaluation of PD(Progressive Disease) or death of any cause.
Antitumor efficacy-Duration of disease control (DDC) | Month 24
  The period from the first evaluation of CR, PR, or SD to the first evaluation of PD or any cause of death.
Antitumor efficacy-Overall survival (OS) | Month 24
  The period from the first infusion to any cause of death
Antitumor efficacy-Objective response rate (ORR); | Month 24
  The number of cases in which tumor size is reduced to PR or CR / the total number of evaluable cases (%). In the event of PR or CR, the subjects should confirm it no less than 4 weeks after the first evaluation
Antitumor efficacy-Disease control rate (DCR) | Month 24
  The number of cases in which response (PR + CR) and stable disease (SD) are achieved from the start of cell infusion/the total number of evaluable cases (%).

CONTACTS AND LOCATIONS:
Overall Officials: Qin shukui, Pro, Principal Investigator — The 81st Hospital of PLA; Zhai bo, Pro, Principal Investigator — RenJi Hospital
Locations (6):
- China (6):
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The 81st Hospital of Chinese PLA, Nanjing, Jiangsu
  - Renji Hospital Shang Hai Jiaotong Unversity of Medicine, Shanghai, Shanghai Municipality
  - Zhongshan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No